CLINICAL TRIAL: NCT06280222
Title: Virtual Reality (VR)-Based Intervention to Improve Pre-operative Anxiety in Patients Undergoing Elective Oocyte Cryopreservation: a Randomized Clinical Trial
Brief Title: The Effectiveness of Virtual Reality on Anxiety Reduction in Women Undergoing Elective Egg Cryopreservation.
Acronym: VRFORANXIETY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, SUISSA COHEN YAEL, Doctor, MD, Principal investigator, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VR FOR ANXIETY-HMO-CTIL
Record Dates: First submitted 2023-12-07; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine management (No Intervention): Usual care of patients prior to a surgical procedure : oocyte retrieval
- Virtual reality management (Experimental): 20 minutes of scenery VR movies prior to the surgical procedure (oocyte retrieval)
  Interventions: Device: The VR instrument - Oculus Quest 2

INTERVENTIONS:
Device: The VR instrument - Oculus Quest 2 — Patients in the interventional group will watch 20-minute scenery movies in the VR instrument before entering the oocyte retrieval procedure.
  Arms: Virtual reality management

SUMMARY:
A randomized trial assessing the effectiveness of virtual reality exposure prior to an oocyte retrieval procedure in terms of anxiety level .

DETAILED DESCRIPTION:
Eligible women, undergoing elective egg freezing, will be offered to participate in the study, and sign a consent form.

The patients will be randomized into 2 groups:

1. No intervention (routine management).
2. Exposure to scenery video, as a VR (virtual reality) session.

All women will be addressed prior to the procedure, while they are waiting, and upon consent will be asked to state their VAS (visual analogue scale) anxiety score and to fill the STAI (The State-Trait Anxiety Inventory questionnaire.) Vital signs (Heart rate, Blood pressure) will be recorded upon arrival.

Patients who were allocated to the VR arm will watch a 20-minute scenery video and following the session before entering the procedure will be asked to rate their VAS score and answer the STAI questionnaire once again. vital signs will be recorded again.

After recovery all women will fill the STAI questionnaire, VAS score and vital signs before they will be discharged.

ELIGIBILITY:
Inclusion Criteria:

* Patients before egg retrieval for social reasons (elective egg freezing)

Exclusion Criteria:

* Use of any medications for pain relief/ anti -anxiety /anti -depressants medication generally or prior to the intervention
* If suffers from any condition that Use of VR is not recommended:

  1. Risk for seizures
  2. Sensitivity to ﬂashing light/motion
  3. Predisposing to nausea/dizziness (vertigo, etc.) Any injury to the eyes/face/neck that would limit the use of the hardware, including blindness.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Vital signs | Up to 8 hours from admission. (Admission, pre-procedural, discharge)
  Blood pressure (systolic+ diastolic levels)
Vital signs | Up to 8 hours from admission. (Admission, pre-procedural, discharge)
  Heart rate (Beats per minute)
VAS (visual-analogue scale) | Up to 8 hours from admission. (Admission, pre-procedural, discharge)
  VAS anxiety score (1-10), Higher levels indicate higher anxiety levels.
State and Trait Anxiety (STAI) Score | Up to 8 hours from admission. (Admission, pre-procedural, discharge)
  The patient's anxiety levels will be assessed using the STAI questionnaire, higher numbers in the questionnaire indicate higher anxiety levels. Levels up to 30 indicate low anxiety, between 30-45 moderate anxiety, more than 46 high anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah mound scopus IVF unit, Jerusalem, Israel

REFERENCES:
- [Derived] Suissa-Cohen Y, Frenkel R, Nevo L, Kam HA, Bentov Y, Godin M, Broder EE, Hizkiyahu R, Lazarovits CA, Beharier O, Klement AH. Virtual reality-based intervention to improve pre-operative anxiety in patients undergoing planned oocyte cryopreservation: a randomized clinical trial. J Assist Reprod Genet. 2025 Sep;42(9):2995-3002. doi: 10.1007/s10815-025-03571-w. Epub 2025 Jul 9. PMID 40632426